CLINICAL TRIAL: NCT04766203
Title: Relative Energy Deficiency in Sport (RED-S) in International and Canadian High Performance Athletes: Prevalence, Health and Performance Implications
Brief Title: Relative Energy Deficiency in Sport Multicenter Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Trent Stellingwerff (Other)
Collaborators: Mitacs (Industry); University of British Columbia (Other)
Responsible Party: Sponsor-Investigator, Trent Stellingwerff, Director of Performance Solutions, Innovation & Research for Canadian Sport Institute Pacific (CSI Pacific) Adjunct Faculty - Exercise Science, Physical & Health Education (EPHE), University of Victoria (UVic), University of Victoria
Organization: University of Victoria (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: RED-S multicenter 2020-22
Record Dates: First submitted 2021-02-16; First posted 2021-02-23 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-06

CONDITIONS: Health, Subjective; Nutrition Disorders; Athletic Injuries; Hormone Disturbance; Exercise-related Amenorrhea; Eating Disorders; Sleep Hygiene; Cardiovascular Abnormalities; Bone Fracture; Bone Loss; Weight Change, Body; Mental Health Wellness 1
MeSH Terms: conditions — Nutrition Disorders; Athletic Injuries; Endocrine System Diseases; Feeding and Eating Disorders; Sleep Hygiene; Cardiovascular Abnormalities; Fractures, Bone; Bone Diseases, Metabolic; Body Weight Changes

STUDY DESIGN:
Intervention Model Description: This study will be comprised of: 1) screening of athletes for symptoms of REDS; and 2) treating athletes diagnosed with REDS with a nutritional intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Global screening of high-performance athletes for REDS (No Intervention): This arm collects data with an online survey to assess prevalence and signs and symptoms of REDS in elite female and male elite and recreational athletes and para-athletes over the age of 15 years across the world.
- Basic screening of Canadian high-performance athletes for REDS (No Intervention): In this study arm, varsity level to elite Canadian athletes and para-athletes will complete a baseline blood sample and potentially (where abnormalities are present) a follow-up 6 months later.
- Advanced screening of Canadian high-performance athletes for REDS (No Intervention): In this study arm, varsity level to elite Canadian athletes and para-athletes will complete a baseline test for bone density (DXA scans), resting metabolic rate and exercise testing. Potentially (where abnormalities are present) a follow-up 6 months later.
- Treatment of Canadian athletes with REDS: a holistic intervention arm (Experimental): In this arm, varsity level to elite Canadian athletes and para-athletes with REDS will participate in a nutritional intervention aiming to improve energy availability and thus, REDS status.
  Interventions: Behavioral: Treatment of REDS using a holistic treatment arm

INTERVENTIONS:
Behavioral: Treatment of REDS using a holistic treatment arm — This arm aims to treat athletes with REDS symptoms by implementing a holistic, individualized nutrition intervention to improve energy availability and thus restore impaired body function due to REDS.
  Arms: Treatment of Canadian athletes with REDS: a holistic intervention arm

SUMMARY:
Relative Energy Deficiency in Sport (RED-S) characterizes a range of negative health and performance outcomes that result from chronically low energy availability. RED-S concerns high performance junior and senior athletes across Canada and has a prevalence rate of 3-60%. Our ability to assess and diagnose RED-S remains poor. Accordingly, we aim to create the best parameters to diagnose and manage RED-S; along with information of the prevalence and severity across Canada and globally. These outcomes are expected to have a significant positive impact on the health and performance of Canadian athletes in preparation for the Olympic Games in 2022 and beyond.

DETAILED DESCRIPTION:
Purpose:

Our aim is to improve our understanding of the prevalence and symptoms of RED-S in international and Canadian athletes and para-athletes, along with developing screening tools and treatment protocols to manage RED-S in order to improve athlete health, availability and performance.

Objectives:

1. Assess the prevalence of self-reported RED-S health outcomes in international and Canadian elite female and male athletes and para-athletes as well as recreational athletes (Study A);
2. Assess the prevalence and severity of measured standard/basic RED-S health outcomes including biomarkers and potential longitudinal (6-mo) tracking of outcomes across the Canadian Olympic and Paralympic Sport Institute Network (COPSI) (Study B);
3. Implement a more advanced assessment, using novel RED-S assessment parameters in a smaller cohort of key athletes, including potential longitudinal tracking over a 6-mo period (Study C);
4. Assess longitudinal changes and the treatment of RED-S symptoms across a 6-month follow-up period in a small cohort of elite Canadian athletes willing to partake in an 'holistic' RED-S treatment intervention arm (Study D);
5. Utilize the data created from Studies A,B,C,and D to develop and validate potentially novel RED-S assessment parameters in order to further validate the 'new' IOC RED-S clinical assessment tool (CAT) version 2 to aid in the diagnosis of RED-S.

Justification:

This study will be the first to systematically assess the prevalence and severity of outcomes of RED-S in a large group of international and Canadian athletes and para-athletes (A), and within the COPSI network (B,C), utilising physiological and performance tests and training metrics for a more holistic assessment of potential outcomes (B,C,). This study will also aim to strengthen the literature regarding to the time-course of changes in these outcomes (B,C,D) and the efficacy of a simple nutritional intervention arm on these changes (D). Finally, this multicentre project will be the largest to date in Canada and globally, and the first to produce data on the prevalence of RED-S within the COPSI network (across A,B,C,D).

Research Design:

This is an observational study including online survey and physiological testing with potential for follow-up in a subset of athletes. A separate study arm (study D) will be an intervention arm with follow-up.

Statistical analysis:

Analysis will be a combination of basic statistics such as t-tests and ANOVA's, as well as more advanced statistical modelling (e.g. stepwise regression modelling, with first identifying collinearity among independent variables via the implementation of variance inflation factors (VIFs)) as well as questionnaire-based statistics and potentially principal components analysis (PCA) will be implemented.

Physiological data will be plotted against survey data to create links between RED-S symptoms among various athlete groups (female vs male, able bodied vs disabled, sports groups, age categories, etc.)

ELIGIBILITY:
Inclusion Criteria:

* International or Canadian elite (National Sport Organization identified) and (Provincial Sport Organization / University varsity identified) Next Generation, or recreational athlete or para-athlete
* Female or male athlete or para-athlete currently and actively training for and racing in an Olympic sports event
* Age >15 years

Exclusion Criteria:

* Under 15 years old
* Pregnant

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
REDS clinical assessment tool and REDS risk score | Baseline and possibly change after 6 months for a subset of athletes
  a combination of validated and semi-validated questionnaires
Menstrual function in females | Baseline and possibly change after 6 months for a subset of athletes
  via Low Energy Availability in Females Questionnaire (higher scores reflect higher risk of RED-S) and use of urinary ovulation strips to measure LH surge
Triiodothyronine concentrations | Baseline and possibly change after 6 months for a subset of athletes
  Venous blood samples
Estrogen concentrations | Baseline and possibly change after 6 months for a subset of athletes
  Venous blood samples
Testosterone concentrations | Baseline and possibly change after 6 months for a subset of athletes
  Venous blood samples
Luteinizing hormone concentrations | Baseline and possibly change after 6 months for a subset of athletes
  Venous blood samples
Follicle-stimulating hormone concentrations | Baseline and possibly change after 6 months for a subset of athletes
  Venous blood samples
Sex-hormone binding globulin concentrations | Baseline and possibly change after 6 months for a subset of athletes
  Venous blood samples
Hemoglobin concentrations | Baseline and possibly change after 6 months for a subset of athletes
  Venous blood samples
Ferritin concentrations | Baseline and possibly change after 6 months for a subset of athletes
  Venous blood samples
Serum iron concentrations | Baseline and possibly change after 6 months for a subset of athletes
  Venous blood samples
Total iron binding capacity | Baseline and possibly change after 6 months for a subset of athletes
  Venous blood samples
Iron saturation | Baseline and possibly change after 6 months for a subset of athletes
  Venous blood samples
Total cholesterol concentrations | Baseline and possibly change after 6 months for a subset of athletes
  Venous blood samples
LDL cholesterol concentrations | Baseline and possibly change after 6 months for a subset of athletes
  Venous blood samples
HDL cholesterol concentrations | Baseline and possibly change after 6 months for a subset of athletes
  Venous blood samples
Triglycerides concentrations | Baseline and possibly change after 6 months for a subset of athletes
  Venous blood samples
Bone mineral density | Baseline
  Dual energy x ray scan of lumbar spine and femoral neck bone density
Resting metabolic rate | Baseline and possibly change after 6 months for a subset of athletes
  Assessment done with a metabolic cart by collecting respiratory gases
Aerobic capacity | Baseline and possibly change after 6 months for a subset of athletes
  maximal oxygen uptake test
Strength | Baseline and possibly change after 6 months for a subset of athletes
  Maximal strength tests
Insulin like growth factor 1 concentrations | Baseline and possibly change after 6 months for a subset of athletes
  Venous blood samples
Resting heart rate | Baseline and possibly change after 6 months for a subset of athletes
  Heart rate monitor (Polar electro)
Blood pressure (systolic and diastolic) | Baseline and possibly change after 6 months for a subset of athletes
  Blood pressure monitor
Bone stress injury history | Baseline and possibly change after 6 months for a subset of athletes
  online questionnaire on type and number of injuries

SECONDARY OUTCOMES:
Body composition | Baseline and possibly change after 6 months for a subset of athletes
  Via DXA or skinfold calipers
Complete blood count | Baseline and possibly change after 6 months for a subset of athletes
  Venous blood samples
Insulin concentrations | Baseline and possibly change after 6 months for a subset of athletes
  Venous blood samples
Glucose concentrations | Baseline and possibly change after 6 months for a subset of athletes
  Venous blood samples
Cortisol concentrations | Baseline and possibly change after 6 months for a subset of athletes
  Venous blood samples
Prolactin concentrations | Baseline and possibly change after 6 months for a subset of athletes
  Venous blood samples
25(OH)D concentrations | Baseline and possibly change after 6 months for a subset of athletes
  Venous blood samples
illness history | Baseline and possibly change after 6 months for a subset of athletes
  online questionnaire on frequency of illness in the past 24 months
Soft-tissue injury history | Baseline and possibly change after 6 months for a subset of athletes
  online questionnaire on the type and number of injuries in the past 24 months
Sleep hygiene | Baseline and possibly change after 6 months for a subset of athletes
  Athlete Sleep Screening Questionnaire (higher scores reflect sleep impairments)
Mental health | Baseline and possibly change after 6 months for a subset of athletes
  Depression, anxiety and stress scale 21 (higher scores reflect increased mental challenges)
Male athlete health | Baseline and possibly change after 6 months for a subset of athletes
  Low Energy Availability in Males Questionnaire (scoring is under development but higher scores reflect higher risk of REDS)
Gut health | Baseline and possibly change after 6 months for a subset of athletes
  Sections from the LEAF-Q (higher scores reflect higher risk of REDS)
Cardiac health | Baseline and possibly change after 6 months for a subset of athletes
  Questions from the Pre-Participation Examination questionnaire (higher scores reflect higher risk of cardiac symptoms)
Mood state | Baseline and possibly change after 6 months for a subset of athletes
  Brunel Mood Scales (higher scores reflect higher mood disturbance)
Eating disorder assessment | Baseline and possibly change after 6 months for a subset of athletes
  Eating Disorder Examination 3 (higher scores reflect higher risk of eating disorders)
History of weight change | Baseline and possibly change after 6 months for a subset of athletes
  online questionnaire
History of anemia | Baseline and possibly change after 6 months for a subset of athletes
  online questionnaire
REDS treatment arm | Individualised but likely 3-6 months
  holistic nutrition based treatment of REDS symptoms including increasing energy availability via nutrition counselling

CONTACTS AND LOCATIONS:
Overall Officials: Trent Stellingwerff, Ph.D., Principal Investigator — Canadian Sport Institute Pacific, University of Victoria, University of British Columbia
Locations (1):
- University of Victoria, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
No data will be shared with researchers outside of the study team.